CLINICAL TRIAL: NCT01721031
Title: Comparison of Dorsal Penile Nerve Block With 0.33% Ropivacaine and Intravenous Tramadol for Prevention of Catheter-related Bladder Discomfort: Study Protocol for a Randomized Controlled Trial
Brief Title: DPNB for Prevention of CRDB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ren Liao, Doctor, Associate professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DPNB120928; LRWCHA (Other: WestChinaH)
Record Dates: First submitted 2012-10-27; First posted 2012-11-02 (Estimated); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Indwelling Urinary Catheter; Male Patients; General Anesthesia
Keywords: Catheter Related Bladder Discomfort; Dorsal Penile Nerve Block
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DPNB (Experimental): Patients receive DPNB 30min before extubation at the end of operation.
  Interventions: Procedure: DPNB
- Tramadol (Active Comparator): Patients receive intravenous tramadol 1.5mg/kg 30min before extubation at the end of operation.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Procedure: DPNB — Patients receive DPNB 30min before extubation at the end of operation
  Arms: DPNB
Drug: Tramadol — Patients receive intravenous tramadol 1.5mg/kg 30min before extubation at the end of operation.
  Arms: Tramadol

SUMMARY:
Catheter-related bladder discomfort (CRBD) secondary to an indwelling urinary catheter is defined as an urge to void or discomfort in the supra-pubic region. This symptom complex may cause patient agitated and exacerbated postoperative pain. In clinic, dorsal penile nerve block (DPNB) was applied for penile surgery including circumcision and some anterior urethra surgery. The investigators hypothesize that DPNB relive CRBD for male patients with indwelling urinary catheter under general anesthesia.

DETAILED DESCRIPTION:
CRBD is not uncommon in the postoperative period, especially in male patients who have had urinary catheterization after anesthetic induction under general anesthesia, and this symptom complex may cause patient agitated and exacerbated postoperative pain. According to the previous study, i.v. tramadol 1.5 mg/kg administered 30 min before extubation results in reduction in the incidence and severity of CRBD. In clinical practice, tramadol is associated with side effects including nausea, vomiting, sedation, etc. Clinically, dorsal penile nerve block (DPNB) was applied in penile surgery, and got satisfactory pain relief effect postoperatively without side effects related to tramadol. Besides, we observed patients underwent urethra surgery with urinary catheter left in situ seldom complained of CRBD if DPNB and RB performed at the end of operation. We hypothesized that DPNB could relieve DPNB for male patient with indwelling urinary catheter insertion after induction of general anesthesia.

In this study we compare the efficacy of dorsal penile nerve block (DPNB) with 0.33% ropivacaine and intravenous tramadol 1.5mg/kg in prevention of CRBD, as well as the incidences of side effects postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed
* Male adult patient, aged 18~50 years old, ASA I~III
* Surgery under general anesthesia

Exclusion Criteria:

* Bladder dysfunction, such as overactive bladder
* A history of bladder outflow obstruction
* Prostate disease, such as benign prostate hyperplasia, etc.
* Disturbance of central nervous system

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-15 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of CRBD | up to 6 months

SECONDARY OUTCOMES:
Visual analogue scale (VAS) for postoperative pain | up to 6 months
Postoperative fentanyl requirement | up to 6 months
Side effects | up to 6 months
  1. the level of sedation.
  2. postoperative nausea vomiting (PONV)
  3. incidence of respiratory depression
  4. incidence of agitation, and delirium

OTHER OUTCOMES:
Acceptance of indwelling urinary catheter | up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Li JY, Yi ML, Liao R. Dorsal Penile Nerve Block With Ropivacaine-Reduced Postoperative Catheter-Related Bladder Discomfort in Male Patients After Emergence of General Anesthesia: A Prospective, Randomized, Controlled Study. Medicine (Baltimore). 2016 Apr;95(15):e3409. doi: 10.1097/MD.0000000000003409. PMID 27082620
- [Derived] Li JY, Liao R. Dorsal penile nerve block with ropivacaine versus intravenous tramadol for the prevention of catheter-related bladder discomfort: study protocol for a randomized controlled trial. Trials. 2015 Dec 30;16:596. doi: 10.1186/s13063-015-1130-2. PMID 26715519